CLINICAL TRIAL: NCT03299114
Title: THE EFFECTIVENESS OF WHIRLPOOL FOR PATIENTS WITH NEUROPATHIC PAIN DUE TO KNEE OSTEOARTHRITIS
Brief Title: WHIRLPOOL FOR OSTEOARHRITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, ASLIHAN UZUNKULAOGLU, Ufuk University, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30112015-6
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Neuropathic Pain; Osteo Arthritis Knee; Sleep Disorder
Keywords: Neuropathic Pain; Whirlpool; Osteoarthritis; Sleep
MeSH Terms: conditions — Neuralgia; Sleep Wake Disorders; Osteoarthritis | interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Treated with warm whirlpool
  Interventions: Other: Whirlpool
- Placebo group (Placebo Comparator): Treated with sham whirlpool
  Interventions: Other: Whirlpool

INTERVENTIONS:
Other: Whirlpool

SUMMARY:
Both neuropathic and nociceptive mechanisms may contribute to the OA pain experience. Aims: The aim of this study was to determine the efficacy of warm whirlpool on pain, disability, quality of life (QoL) and sleep for patients with neuropathic pain.

DETAILED DESCRIPTION:
Whirlpool treatment method is used for medical and surgical conditions. In literature there are studies which recommend whirlpool therapy as a treatment for reducing pain in patients with osteoarthritis. The aim of this study was to determine the efficacy of warm whirlpool on pain, disability, quality of life (QoL) and sleep for patients with neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* suffering from knee pain at least 3 months
* radiological manifestations considering were consistent with grade 3 and 4 knee OA due to Kellgren and Lawrence criteria had DN4 scores ≥4.

Exclusion Criteria:

* lower extremity surgery history, knee infection inflammatory disease like rheumatoid arthritis back or pelvic pain related with knee pain another cause of polyneuropathy (diabetes mellitus, vitamin B 12 deficiency, toxic or neurological disease like stroke, spinal cord injury) lumbar disc herniation malignancy or active systemic disease.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | one month

SECONDARY OUTCOMES:
Short Form-36 Health Survey | one month
Western Ontario and McMaster Universities Osteoarthritis Index | one month
Pittsburgh Sleep Quality Index (PSQI) | one month
DN4 | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No